CLINICAL TRIAL: NCT04745754
Title: The EPICS (Engaging Primary Care in Cancer Survivorship) Study: A Trial of Novel Models of Care for Cancer Survivors
Brief Title: The Engaging Primary Care in Cancer Survivorship (EPICS) Study
Acronym: EPICS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erin E. Hahn, Research Scientist I, Kaiser Permanente
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA249419 (NIH); 1R01CA249419-01 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Cancer survivorship; Models of care
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Embedded primary care providers (PCPs) will provide comprehensive care for survivors, including cancer surveillance services, preventive care, and management of long-term therapy and associated side effects (e.g., endocrine therapy in breast survivors). A comprehensive multilevel approach will prepare survivors and PCPs (physicians and/or advance practice providers). Eligible patients in the embedded PCP model will be provided with tailored education regarding the planned transition and, after cessation of active treatment, printed information on the planned course of care, expectations for embedded PCP care, transition timing, and reassurance that the oncology team will be available via telephone and email, and that PCPs will refer back to the oncologist for any concerning signs or symptoms. Tailored alerts will also be added to the electronic medical record (EMR) for recommended cancer surveillance and preventive care services that will fire for visits with embedded PCPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): The trial will test the efficacy of an embedded primary care provider (PCP) model (experimental condition) in which PCPs are trained in survivorship and then embedded within an oncology practice to care for low-risk, early stage breast and colorectal cancer survivors who will be transitioned at 6-36 months post-treatment for comprehensive survivorship care.
  Interventions: Other: Embedded primary care in cancer survivorship model
- Control Condition (No Intervention): Usual care for breast and colorectal cancer survivors (oncology-led model).

INTERVENTIONS:
Other: Embedded primary care in cancer survivorship model — Primacy care physicians will receive comprehensive training in cancer survivorship care for low-risk, early stage breast and colorectal patients. Training will include continuing medical education (CME) modules, webinars, and in-person discussion and clinical shadowing.
  Arms: Intervention Condition

SUMMARY:
A quasi-experimental non-randomized pre/post with control group trial of two models of cancer survivorship care in early-stage colorectal and breast cancer survivors cared for in a community-based, integrated health care setting.

DETAILED DESCRIPTION:
A quasi-experimental non-randomized pre/post with control group trial of two models of cancer survivorship care in early-stage colorectal and breast cancer survivors cared for in a community-based, integrated health care setting. The trial will test the efficacy of an embedded primary care provider (PCP) model (experimental condition) in which PCPs are embedded within an oncology practice and will care for low-risk survivors who will be transitioned at 6-36 months post-treatment for comprehensive survivorship care. We hypothesize that a) patients in the PCP model will have superior receipt of recommended care compared to usual care; b) patients in the PCP model will perceive significantly better care coordination, self-efficacy, and confidence in their PCP compared to usual care; and c) use of unplanned and non-recommended care will be less in the PCP model compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Adult (21+) Kaiser Permanente Southern California members diagnosed and treated for pathologically confirmed first primary early-stage breast (stage 0, I, II) or colorectal (stage I, II) cancer within Kaiser Permanente Southern California. Completed active cancer treatment within the past 6-36 months; active treatment includes cancer-directed surgery, chemotherapy (includes Herceptin (Trastuzumab)), radiation therapy, and ovarian suppression therapy (e.g., Goserelin (Zoladex)). Completed at least one office visit within Kaiser Permanente Southern California medical oncology. At low-risk for cancer recurrence and treatment-related toxicities based on state of disease and treatment modalities. For our Aim 2 survey: Primary language of English or Spanish (although we will assess our Aim 1 participants for recorded preferred spoken language and adjust translations as needed). Ability to complete surveys of patient-reported outcomes.
* Physicians: For centers assigned to the embedded primary care physician (PCP) model, PCPs selected to participate must be Board Certified in a relevant primary care specialty; hold a valid and current MD or advanced practitioner license; and be employed by the Southern California Permanente Medical Group.

Exclusion criteria:

* Patients less than 21 years of age
* Patients at high risk for recurrence and treatment-related toxicities based on stage of disease and treatment modalities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2450 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cancer surveillance care services | 36 months
  Receipt of guideline-recommended cancer surveillance care services.
Preventive care services | 36 months
  Receipt of guideline-recommended preventive care services.

SECONDARY OUTCOMES:
Non-recommended surveillance care/non-planned emergency and urgent care services | 36 months
  Receipt of non-recommended surveillance care based on current clinical guidelines, and use of non-planned hospitalization, emergency department, and urgent care services.
Medical Expenditure Panel Survey (MEPS) 2016, Experiences with Cancer Supplement, Section 7, Medical Care for Cancer Module (Item #44) | 12 months
  Validated measures of cancer survivorship financial burden, access to medical care, employment and employment patterns, healthcare utilization and expenditures, and use of prescription drugs by cancer survivors (Item #44; response options: 4-item Likert scale)
Patient-Centered Medical Home (PCMH) and Cancer Consumer Assessment of Healthcare Providers and Systems (CAHPS) | 12 months
  The Patient-Centered Medical Home (PCMH) Item Set is a set of supplemental questions that can be added to the adult and child versions of the CAHPS Clinician & Group Survey (CG-CAHPS) to gather more information on patient experience with the domains of primary care that define a medical home. However, use of this item set is not limited to practices that explicitly function as medical homes. Any primary care practice that is interested in a more comprehensive assessment of their patients' experiences may add the PCMH items to the survey (6 questions; response options: 3-item, 4-item or 6-item Likert scale).
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2 (answer responses using a Likert Scale) | 12 months
  As part of the Patient-Reported Outcomes Measurement Information System (PROMIS) created in 2004, The PROMIS Global-10 is a publically available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions (10 questions; response options: 5-item Likert scale).
Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions Symptoms Scale (Self-efficacy for managing symptoms short form 8a (8 questions; 5-item Likert scale) | 12 months
  The PROMIS adult Self-Efficacy for Managing Chronic Conditions Symptoms Scale assesses self-reported current level of confidence in managing symptoms from chronic health conditions (8 questions; response options: 5-item Likert scale).
The European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (version 3) | 12 months
  Questionnaire developed to assess the quality of life of cancer patients (30 questions; response options: 4-item or 7-item Likert scale)
Receipt of Treatment Summary from Health Information and National Trends Survey (HINTS 4, Cycle 2) | 12 months
  The Health Information National Trends Survey (HINTS) regularly collects nationally representative data about the American public's knowledge of, attitudes toward, and use of cancer- and health-related information (1 question; response option: yes/no).
Primary Care Delivery of Survivorship Care Scale | 12 months
  Self-reported measure of perceived survivorship care (6 questions; response options: 5-item Likert scale)
Patient-Reported Bother from Side Effects of Cancer Therapy (Validated Single-Item Measure) | 12 months
  The single item "I am bothered by side effects of treatment" (GP5), rated on a 5-point Likert scale, is part of the Functional Assessment of Cancer Therapy-General (FACT-G) version (1 question; response option: 5-item Likert scale)
The Satisfaction with Decision Scale | 12 months
  (6 questions; response options: 4-item Likert Scale)
Confidence in Managing Survivorship Care | 12 months
  Questionnaire assessing self-reported receipt of survivorship care planning, expectations of their providers, and confidence in managing their survivorship care (5 questions; response options: 4-item Likert scales).
Cancer recurrence | 12 months
  Single item, question: Did a doctor or other health professional ever tell you that your cancer had come back? (response option: yes/no). 1a. If yes, what was the most recent year a doctor or other health professional told you that your cancer had come back? _______________

OTHER OUTCOMES:
Self-reported patient demographics | 12 months
  gender, race/ethnicity; insurance type; highest level education; school/employment status; total household income

CONTACTS AND LOCATIONS:
Overall Officials: Erin E. Hahn, PhD, MPH, Principal Investigator — Kaiser Permanente Southern California, Department of Research & Evaluation
Locations (13):
- United States (13):
  - Kaiser Permanente Orange County Anaheim/Irvine Medical Center Oncology Clinics, Anaheim, California
  - Kaiser Permanente Baldwin Park Medical Center Oncology Clinic, Baldwin Park, California
  - Kaiser Permanente Downey/Bellflower Medical Center Oncology Clinics, Downey, California
  - Kaiser Permanente Fontana Medical Center Oncology Clinic, Fontana, California
  - Kaiser Permanente South Bay Medical Center Oncology Clinic, Harbor City, California
  - Kaiser Permanente Kern County Medical Facilities Oncology Clinic, Kern, California
  - Kaiser Permanente Antelope Valley Medical Center Oncology Clinic, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center Oncology Clinic, Los Angeles, California
  - Kaiser Permanente West Lost Angeles Medical Center Oncology Clinic, Los Angeles, California
  - Kaiser Permanente Panorama City Medical Center Oncology Clinic, Panorama City, California
  - Kaiser Permanente Riverside/Palm Springs Medical Center Oncology Clinics, Riverside, California
  - Kaiser Permanente San Diego Medical Center Oncology Clinics, San Diego, California
  - Kaiser Permanente Woodland Hills Medical Center Oncology Clinic, Woodland Hills, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04745754/Prot_SAP_003.pdf